CLINICAL TRIAL: NCT05178550
Title: An Open-label, Randomized, Single Center, Crossover Study in Healthy Participants to Assess Lipoprotein Lipase Activity and Levels, and Triglyceride Levels After Heparin Exposure, in Both Fasted and Postprandial State
Brief Title: A Study in Healthy Participants Investigating Biomarkers After Exposure to Heparin When Heparin is Administered in the Fasted State or After a High-fat Meal. Heparin, a Registered Drug, is an Anticoagulant (Blood Thinner) That Prevents the Formation of Blood Clots.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NN6633-4955; 2021-005899-18 (EudraCT Number); U1111-1270-0957 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-12-14; First posted 2022-01-05 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (low dose-high dose) (Experimental): Participants receive 25 IU/kg heparin on days 1 and 2, and 50 IU/kg Heparin on days 4 and 5
  Interventions: Drug: Heparin
- Group 2 (high dose-low dose) (Experimental): Participants receive 50 IU/kg heparin on days 1 and 2, and 25 IU/kg Heparin on days 4 and 5
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — intravenous [iv] injection

SUMMARY:
In this study biomarkers in the blood after exposure to heparin in the fasted state or after a high-fat meal will be investigated. Heparin will be administered as an intravenous (iv) injection (injection directly in a blood vessel). In this study, the effects of administration of heparin will be compared with the effects of administration of normal saline which will also be administered as an iv injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Male or female
* 18 to 65 years, inclusive, at the time of signing informed consent
* Body mass index:18.0 kg/m ^2 to 29.9 kg/m^2, inclusive, at the time of signing informed consent
* Body weight greater than or equal to 50 kg at the time of signing informed consent

Exclusion criteria:

* Using tobacco products within 60 days prior to the first drug administration.
* Any kind of coagulation disorder or any first degree family members with major bleeding tendency.
* History of anemia, thrombocytopenia, HIT, other blood disorders, or any clinically relevant bleeding (epistaxis).
* Exposure to heparin (unfractionated heparin or low molecular weight heparin) within 100 days prior to the first dose of heparin.
* Participation in any clinical study of an approved or non-approved investigational medicinal product within 30 days (or 5 half-lives of the investigational medicinal product, whichever is greater) before screening. If the half-life of the investigational medicinal product is unknown, subjects participating in a clinical trial in the 6 months prior to (the first) treatment administration will be excluded.
* Any kind of coagulation disorder or any first degree family members with major bleeding tendency.
* Unwillingness to consume the entire high-fat standardized meal (e.g. vegetarians, vegans and subjects who follow special diets).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Lipoprotein Lipase (LPL) levels before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  ng/ml
Change from baseline in LPL activity before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  µmol/l/min
Change from baseline in Triglycerides (TG) levels before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  mmol/L

SECONDARY OUTCOMES:
Change from baseline in apolipoprotein CII (APOCII) levels before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  mg/L
Change from baseline in APOCIII levels before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  mg/dl
Change from baseline in total cholesterol levels before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  mmol/L
Change from baseline in Free fatty acids (FFA) levels before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  mmol/L
Change from baseline in Lipoprotein profiling (very-low-density lipoprotein (VLDL), low-density lipoprotein (LDL), high-density lipoprotein (HDL) before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  mmol.L-1
Change from baseline in adverse events (AEs) before and after heparin exposure both in fasted and postprandial state | day -1 to day 6
  Number of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com